CLINICAL TRIAL: NCT00350662
Title: Randomized Open-label Phase III Study With Deferiprone and/or Desferrioxamine in Iron Overloaded Patients
Brief Title: Study With Deferiprone and/or Desferrioxamine in Iron Overloaded Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lipomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DF-1
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Hemochromatosis
Keywords: Deferiprone; L1; Desferrioxamine; Hemochromatosis; Iron overload; Thalassemia
MeSH Terms: conditions — Hemochromatosis; Iron Overload; Thalassemia | interventions — Deferiprone; Long Interspersed Nucleotide Elements; Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Deferiprone + Desferrioxamine (Experimental)
  Interventions: Drug: Deferiprone (L1); Drug: Desferrioxamine
- Deferiprone single agent (Experimental)
  Interventions: Drug: Deferiprone (L1)
- Desferrioxamine single agent (Active Comparator)
  Interventions: Drug: Desferrioxamine

INTERVENTIONS:
Drug: Deferiprone (L1) — 75 mg/kg body weight daily
  Arms: Deferiprone + Desferrioxamine; Deferiprone single agent
Drug: Desferrioxamine — In combination with deferiprone: 40-50 mg/kg body weight 2-times weekly As single agent: 40-50 mg/kg body weight 5- to 7-times weekly
  Arms: Deferiprone + Desferrioxamine; Desferrioxamine single agent

SUMMARY:
Comparison of efficacy and toxicity of the combination treatment of deferiprone and desferrioxamine with the single agent treatment of either drug

DETAILED DESCRIPTION:
Patients with refractory anemias requiring regular blood transfusions accumulate iron at the rate of approximately 0.5 mg/kg/day, which may lead to serious organ toxicity. The human body has no active mechanism for the excretion of excess iron. Therefore multiply transfused patients will develop a secondary hemosiderosis, if no iron excretion is achieved by a chelating agent. Symptoms of iron-overload occur when body iron stores reach 10-20 g. At higher levels severe, even fatal complications, particularly cardiac failure, may develop.

Desferrioxamine (DFO, Desferal) is the established and commonly used iron-chelating drug, but is expensive and must be given by slow subcutaneous or intravenous infusion for 8-12 hours a day during 5-7 days weekly at a dosage of 40-50mg/kg body weight/day. This often leads to failure of compliance of the patient and therefore to inefficient iron chelation. Further some patients are hypersensitive to desferrioxamine and others suffer from toxicity, e.g. to the ears or eyes.

Deferiprone (L1; CP20; 1,2 dimethyl-3-hydroxy-pyrid-4-one) is an orally active iron chelator investigated in various clinical trials since 1987. Dosages of 75 - 100mg/kg body weight/day of L1 have been found effective to maintain stable iron balance (urinary iron excretion of 0.5mg/kg/day) and to reduce serum ferritin levels between 6% and 25% within one year of treatment in iron-overloaded thalassemic patients. There exists long-term experience with patients who have received deferiprone continuously for more than 10 years so far. However, only few controlled comparison studies with L1 and DFO have been performed so far in order to confirm the effectiveness of deferiprone.

The main side effects encountered during a deferiprone therapy are arthropathy, gastrointestinal symptoms, headache, and mild zinc deficiency. These adverse effects are usually reversed on reducing the dose or discontinuing the drug. Except for severe joint symptoms in few patients, most of the subjects in different clinical trials have been able to continue with L1 therapy for a long-term. The most severe and rare complication following L1 administration is agranulocytosis or neutropenia.

A new treatment regimen by combining deferiprone with desferrioxamine is currently being investigated in many countries. Preliminary data could demonstrate that the combined use of both drugs is highly active showing a synergistic or even additive effect (significant decrease of serum ferritin and hepatic iron content, increase of urinary iron excretion). This synergism could be explained by the different mode of activity of the two drugs. It could be demonstrated that patients who were not sufficiently chelated with desferrioxamine or deferiprone, could achieve a negative iron balance with the combination treatment of both drugs. The combined regimen was generally well-tolerated and there is evidence that the individual toxicity profile of both drugs can be positively influenced by the simultaneous administration of L1 and DFO. The daily treatment with L1 tablets combined with a twice a week administration of parenteral desferrioxamine is more patient-convenient and therefore may enhance the compliance of the patient. In addition, this new treatment regimen will reduce the overall therapy expenses if compared to the high Desferal and material costs related to the parenteral administration of DFO on 5 to 7 days per week.

The results of the previous studies with deferiprone are often not comparable, e.g. laboratory parameters, toxicities and side effects vary from study to study. The number of patients included in the clinical investigations was in general too low to allow statistically significant evaluations. Further, there is no controlled randomized study comprising an appropriate number of patients in order to allow a comparison between the combination arm and the single agent control arms. This study protocol aims to evaluate the feasibility of the combination treatment by comparing the efficacy and safety of the combined drugs with the single agent treatment of L1 and DFO in iron-overloaded patients with thalassemia or refractory anemia in a controlled randomized multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Iron-overloaded patients without prior iron chelation therapy as well as pretreated patients
* Age: 4 years and older
* Sex: male and female
* Written informed consent

Exclusion Criteria:

* Children < 4 years of age
* Patients non-compliant to DFO or L1
* Patients with known DFO or L1 toxicity/intolerance
* Neutropenia (neutrophils < 1.5 x 10exp9/L)
* Thrombocytopenia (platelets < 100 x 10exp9/L)
* Renal, hepatic (liver enzymes 2.5x of upper normal level and higher) or decompensated heart failure
* Active viral illness currently treated with interferon-alpha/ribavirin
* Patients with repeated Yersinia infections
* HIV-positivity
* Pregnancy and nursing
* Female and male of reproductive age planning for family, sexually active but not taking adequate contraceptive precaution

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2002-01

PRIMARY OUTCOMES:
Clinical efficacy (Iron balance and liver iron concentration) | At baseline and at 12 months

SECONDARY OUTCOMES:
Safety profile (general, hematologic, and organ toxicity) | At 3-monthly intervals
Liver histology | At baseline and at 12 months
Quality of life (patient's subjective of compliance and tolerance) | At 3-monthly intervals
Actual treatment duration (ATD) | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Amal M El-Beshlawy, Prof. Dr., Principal Investigator — Pediatric Hospital, Cairo University, Cairo, Egypt; Yesim Aydinok, Prof. Dr., Principal Investigator — EGE University Medical School Bornova, Izmir, Turkey
Locations (2):
- Pediatric Hospital, Cairo University, Cairo, Egypt
- EGE University Medical School, Bornova, Izmir, İzmir, Turkey (Türkiye)

REFERENCES:
- [Result] El-Beshlawy A, Manz C, Naja M, Eltagui M, Tarabishi C, Youssry I, Sobh H, Hamdy M, Sharaf I, Mostafa A, Shaker O, Hoffbrand AV, Taher A. Iron chelation in thalassemia: combined or monotherapy? The Egyptian experience. Ann Hematol. 2008 Jul;87(7):545-50. doi: 10.1007/s00277-008-0471-2. Epub 2008 Mar 20. PMID 18351337
- [Result] Aydinok Y, Ulger Z, Nart D, Terzi A, Cetiner N, Ellis G, Zimmermann A, Manz C. A randomized controlled 1-year study of daily deferiprone plus twice weekly desferrioxamine compared with daily deferiprone monotherapy in patients with thalassemia major. Haematologica. 2007 Dec;92(12):1599-606. doi: 10.3324/haematol.11414. PMID 18055982
- [Result] Aydinok Y, Evans P, Manz CY, Porter JB. Timed non-transferrin bound iron determinations probe the origin of chelatable iron pools during deferiprone regimens and predict chelation response. Haematologica. 2012 Jun;97(6):835-41. doi: 10.3324/haematol.2011.056317. Epub 2011 Dec 16. PMID 22180427